CLINICAL TRIAL: NCT01190605
Title: Evaluating Factors That Impact Loss to Follow-up Among Postpartum HIV-infected Women in Mississippi
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Binford Nash, Asst. Professor, Pediatrics, School of Medicine, University of Mississippi Medical Center
Other Study IDs: 2010-0131
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: HIV
Keywords: HIV; postpartum; postpartum entry into HIV care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Women with HIV infection in Mississippi who are pregnant or who have had their baby in the past year can agree to fill out a questionnaire about what helps or hurts return to care for HIV infection after having a baby. The combined results should show the most common things that keep women from getting care for HIV infection after having a baby. This will help design another study in order to help more women get into care for HIV infection after having a baby.

DETAILED DESCRIPTION:
Following recruitment and completion of informed consent, a participant will be given a questionnaire to look at factors that help or hinder access to HIV care after delivery. After finishing the initial questionnaire the participant will get a Wal-Mart gift card for $15. The participant may then be asked to complete a longer interview for which she would receive an additional gift card for $25. The combined results will be used to design an interventional study to improve entry into HIV care after delivery.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* women with HIV infection who are pregnant or up to 2 months postpartum
* English speaking
* able to give informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women in Mississippi with HIV infection who have been pregnant and received perinatal HIV care at University of Mississippi Medical Center are eligible to participate in a questionnaire study on the factors that affect entry into HIV care after delivery
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
linked to long-term HIV care | within six months of delivery
  retrospective chart review for documentation of visit attendance

SECONDARY OUTCOMES:
assessment for depression | cross-sectional at time of study visit
  use of Edinburgh depression screening tool
assessment of intimate partner violence | cross-sectional at time of study visit
  use of WEB (Women's Experience with Battering) screening tool
assessment of stigma | cross-sectional at time of study visit
  use of HIV Related Experiences screening tool
attended a postpartum visit | within six months of delivery
  retrospective chart review for documentation of visit attendance

CONTACTS AND LOCATIONS:
Overall Officials: Binford T Nash, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States